CLINICAL TRIAL: NCT06033261
Title: A Phase 1/2, Randomized, Observer-Blind, Controlled, Dose-Ranging Study of mRNA-1608, an HSV-2 Therapeutic Candidate Vaccine, in Healthy Adults 18 to 55 Years of Age With Recurrent HSV-2 Genital Herpes
Brief Title: A Study of mRNA-1608, a Herpes Simplex Virus -2 (HSV-2) Therapeutic Candidate Vaccine, in Healthy Adults 18 to 55 Years of Age With Recurrent HSV-2 Genital Herpes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mRNA-1608-P101
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Genital Herpes
Keywords: HSV-2; Herpes Simplex Virus Type 2; HSV-2 vaccine; Genital Herpes; mRNA-1608
MeSH Terms: conditions — Herpes Genitalis | interventions — 4CMenB vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- mRNA-1608 Dose A (Experimental): Participants will receive 2 intramuscular (IM) injections of mRNA-1608 at Dose Level A, each dose administered at 0 and 2 months (Day 1 and Day 57).
  Interventions: Biological: mRNA-1608
- mRNA-1608 Dose B (Experimental): Participants will receive 2 IM injections of mRNA-1608 at Dose Level B, each dose administered at 0 and 2 months (Day 1 and Day 57).
  Interventions: Biological: mRNA-1608
- mRNA-1608 Dose C (Experimental): Participants will receive 2 IM injections of mRNA-1608 at Dose Level C, each dose administered at 0 and 2 months (Day 1 and Day 57).
  Interventions: Biological: mRNA-1608
- BEXSERO (Other): Participants will receive 2 IM injections of BEXSERO, each dose administered at 0 and 2 months (Day 1 and Day 57).
  Interventions: Biological: BEXSERO

INTERVENTIONS:
Biological: mRNA-1608 — Sterile liquid for injection
  Arms: mRNA-1608 Dose A; mRNA-1608 Dose B; mRNA-1608 Dose C
Biological: BEXSERO — A vaccine indicated for active immunization to prevent invasive disease caused by Neisseria meningitidis serogroup B.
  Arms: BEXSERO

SUMMARY:
The purpose of this study is to generate safety and immunogenicity data and establish a proof-of-concept of clinical benefit of the mRNA-1608 vaccine candidate.

DETAILED DESCRIPTION:
Participants with a history of recurrent genital herpes will be randomly assigned in a 1:1:1:1 ratio to receive mRNA-1608 at 1 of the 3 dose levels or control (BEXSERO) administered as 2 doses at 0 and 2 months (Day 1 and Day 57).

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of genital HSV-2 infection for at least 1 year before the Screening Visit.
* Seropositive for HSV-2 as determined by Western Blot.
* Participant has a history of recurrent genital herpes defined as at least 3 and no more than 9 reported genital herpes recurrences in the 12 months preceding the Screening Visit, or if currently on suppressive therapy, prior to initiation of suppressive therapy.
* Willing to refrain from taking suppressive antiviral therapy from the Screening Visit until the end of the study.
* Willing to refrain from the use of episodic antiviral therapy during the three 28-day anogenital swabbing periods. Episodic therapy may be used outside the three 28-day swabbing periods.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception, and not currently breastfeeding.

Exclusion Criteria:

* Prior immunization with a vaccine containing HSV antigens.
* History of any form of ocular HSV infection, HSV-related erythema multiforme, or HSV-related neurological complications.
* History of genital HSV-1 infection.
* History of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) types 1 or 2 (HIV-1, HIV-2).
* Reported history of anaphylaxis or severe hypersensitivity reaction after receipt of any mRNA vaccine(s) or any components of the mRNA vaccines.
* Previously received BEXSERO or other vaccine to prevent serogroup B meningococcal disease (also known as meningitis B).
* History of allergic disease or reactions likely to be exacerbated by any component of BEXSERO vaccine.
* Has received or plans to receive any licensed or authorized vaccine, including COVID-19 vaccines, ≤ 28 days prior to the first study injection (Day 1), or plans to receive a licensed or authorized vaccine within 28 days before or after study injection with the exception of licensed influenza vaccines, which may be received more than 14 days before or after any study injection.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 365 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) | Up to Day 64 (7 days after each injection)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 85 (28 days after each injection)
Number of Participants with Serious Adverse Events (SAEs) | Day 1 to Day 393 (end of study [EoS])
Number of Participants with Adverse Events of Special Interest (AESIs) | Day 1 to Day 393 (EoS)
Number of Participants with AEs Leading to Discontinuation From Study | Day 1 to Day 393 (EoS)
Number of Participants with Medically-Attended AEs (MAAEs) | Day 1 through 6 months after last study injection (Day 225)

SECONDARY OUTCOMES:
Number of Genital Herpes Recurrences, Counted Starting 14 Days After the Second Study Injection to 6 Months After Second Study Injection | Day 71 to Day 225
Number of Genital Herpes Recurrences, Counted Starting 14 Days After the Second Study Injection to 12 Months After Second Study Injection | Day 71 to Day 393
Change From Baseline (28 Days Prior to the First Study Injection) to 2 Months After the Second Study Injection in Genital Herpes Lesion Rate (Proportion of Days With Lesions Present) | Baseline (Day -27 to Day 1), Day 85 to Day 113
  To calculate the 'Change from Baseline', the herpes lesion rate during the timeframe of Day 85 to Day 113 will be compared against the herpes lesion rate during the timeframe of Day -27 to Day 1 (Baseline).
Change From Baseline (28 Days Prior to the First Study Injection) to 6 Months After the Second Study Injection in Genital Herpes Lesion Rate (Proportion of Days With Lesions Present) | Baseline (Day -27 to Day 1), Day 197 to Day 225
  To calculate the 'Change from Baseline', the herpes lesion rate during the timeframe of Day 197 to Day 225 will be compared against the herpes lesion rate during the timeframe of Day -27 to Day 1 (Baseline).
Change From Baseline (28 Days Prior to the First Study Injection) to 2 Months After the Second Study Injection in HSV-2 Genital Shedding Rate (Proportion of HSV-2 Deoxyribonucleic acid [DNA] Positive Anogenital Swabs) | Baseline (Day -27 to Day 1), Day 85 to Day 113
  To calculate the 'Change from Baseline', the HSV-2 genital shedding rate during the timeframe of Day 85 to Day 113 will be compared against the HSV-2 genital shedding rate during the timeframe of Day -27 to Day 1 (Baseline).
Change From Baseline (28 Days Prior to the First Study Injection) to 6 Months After the Second Study Injection in HSV-2 Genital Shedding Rate (Proportion of HSV-2 DNA Positive Anogenital Swabs) | Baseline (Day -27 to Day 1), Day 197 to Day 225
  To calculate the 'Change from Baseline', the HSV-2 genital shedding rate during the timeframe of Day 197 to Day 225 will be compared against the HSV-2 genital shedding rate during the timeframe of Day -27 to Day 1 (Baseline).
Geometric Mean Titer (GMT) of mRNA-1608 Antigen-Specific Binding Antibodies (bAbs) at 1 and 6 Months After the Second Study Injection | Days 85 and 225
Geometric Mean Fold Rise (GMFR) of mRNA-1608 Antigen-Specific bAbs From Baseline to 1 and 6 Months After the Second Study Injection | Baseline (Day 1), Days 85 and 225
Number of Participants With Vaccine Seroresponse | Baseline (Day 1), Days 85 and 225
  Seroresponse is defined by an increase in HSV-2 bAb levels at Day 85 and Day 225 ≥4-fold if baseline level is above the lower level of quantitation (LLOQ) or ≥4 × LLOQ if baseline bAb level is <LLOQ prior to study injection.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Accel Clinical Sites Network - Cahaba Medical Care, Birmingham, Alabama
  - Noble Clinical Research, Tucson, Arizona
  - Cedars-Sinai Medical Center/Carbon Health, Beverly Hills, California
  - Acclaim Clinical Research, San Diego, California
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Johnson County Clin-Trials (JCCT), Lenexa, Kansas
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Research Works, New Orleans, Louisiana
  - Fenway Health, Boston, Massachusetts
  - DM Clinical Research, Southfield, Michigan
  - Velocity Clinical Research, Grand Island, Nebraska
  - Velocity Clinical Research, Norfolk, Nebraska
  - Rochester Clinical Research, Rochester, New York
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Velocity Clinical Research Cleveland, Beachwood, Ohio
  - Velocity Clinical Research, Austin, Cedar Park, Texas
  - Helios CR, Inc Fort Worth, Fort Worth, Texas
  - DM Clinical Research, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Health Research of Hampton Roads, Newport News, Virginia
  - University of Washington Virology Research Clinic, Seattle, Washington